CLINICAL TRIAL: NCT03996941
Title: Harm Reduction Program For Informal PrEP Users In A Community-based Setting
Brief Title: Harm Reduction Program For Informal PrEP Users In A Community-based Setting (seguiPrEP)
Acronym: seguiPrEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BCN Checkpoint (Industry)
Collaborators: Projecte dels NOMS Hispanosida (Other); Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Other Study IDs: BCP-FTD-2019-01
Record Dates: First submitted 2019-06-17; First posted 2019-06-25 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: HIV/AIDS; HIV Infections; Sexually Transmitted Diseases; Vaccination; Adherence, Medication; Side Effect of Drug; Preexposure Prophylaxis
Keywords: PrEP; Community setting; point of care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Sexually Transmitted Diseases; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- seguiPrEP: MSM and TGW using or willing to use PrEP informally will be followed in a prospective cohort to describe safety and efficacy, and to provide them with the necessary clinical controls for using it in a safe manner.
  Interventions: Behavioral: Harm reduction of informal PrEP use; Other: PrEP follow up based on point of care testing

INTERVENTIONS:
Behavioral: Harm reduction of informal PrEP use — Users attending the study center interested in PrEP use , as well as those who could benefit from it are invited to attend an information session in which issues are touched like the effectiveness and safety of PrEP, and the characteristics of the SeguiPrEP program. This program consists of periodic clinical controls (five during the first year and four in the following period) that include: physical examination, HIV and other STI screening, control of renal functions, estimation and promotion of PrEP adherence, monitoring of adverse events associated with PrEP and counseling.
  Those who decide to use PrEP or who are already using PrEP are asked to schedule an initiation visit.
Other: PrEP follow up based on point of care testing — The study center has a point-of-care technology based laboratory, which allows obtaining immediate results in order to reduce the loss of follow-up.

SUMMARY:
Pre-Exposure Prophylaxis (PrEP) is a biomedical strategy consisting of the use of antiretroviral therapy by HIV-seronegative people at high risk of acquiring HIV, to prevent the infection. Many controlled and randomized clinical trials, as well as implementation projects have shown that the use of tenofovir disoproxil (TDF) and emtricitabine (FTC) is both safe and effective in the prevention of HIV infection.

However, the administrative situation of PrEP in Spain is anomalous. Unlike in some European countries, PrEP is not available within the National Health System (SNS), although being available for the treatment of HIV infection. In Spain the fixed-dose combination of FTC / TDF is for hospital use only, which requires prescription by HIV specialists exclusively and restricts its dispensation to pharmacy services within the hospital.

This limitation in access and the knowledge of its prevention capacity of PrEP by vulnerable population has led them to obtain "generic FTC / TDF" outside the standardized health care system. According to a survey conducted in Europe to characterize MSM users of PrEP carried out in 2016, 5% of PrEP users had acquired it on their own. Of these 70% stated they were not included in any regular follow-up program while using the medication. Despite the growing demand, there are no health programs (including information, counseling, systematic screening for sexually transmissible infection (STI), etc.) aimed at meeting the health care needs of those who already use or wish to use PrEP, neither by public nor private healthcare providers. This type of service is especially necessary when considering that, among PrEP users, one may have already an established HIV infection, theoretical increase of other STI and a lack of monitoring kidney functions..

BCN Checkpoint is a community center since 2006 for the detection of HIV and other STI aimed at gay men, other men who have sex with men (MSM) and transgender women (TGW), which has shown high efficiency in HIV screening and fast referral to standard HIV care and treatment.. In 2017 the organization opened BCN PrEP·Point, a community centre with the goal to provide information, to conduct clinical trials and clinical monitoring of informal PrEP use.

For this reason, it is presented here the protocol of the SeguiPrEP study, prospective, longitudinal study of health care in the community environment, to MSM and TGW, users of informal PrEP, based on point-of-care testing technology.

DETAILED DESCRIPTION:
In Catalonia 62% of new HIV diagnoses were reported in MSM in 2017. In the decade 2007-2016 in this population group an increase in the number of HIV cases of approximately 44%. The knowledge, interest and willingness to use PrEP is high among MSM at higher risk of HIV acquisition. BCN Checkpoint was accountable for the detection of one third of all new HIV cases in MSM and TGW in Catalonia.

Research hypothesis is that offering a risk reduction program, including the provision of health monitoring, in a community setting for informal PrEP users is justified and feasible, and will afford these users the possibility of using it safely. It is expected that the use of informal PrEP, along with HIV and other STIs screening, STI treatment, and immediate HIV referral to care and treatment will contribute significantly to a reduction of HIV incidence.

This study aims to contribute to increase the body of evidence on the incidence and of context specific HIV management and inform policy makers on potential preventive strategies against the epidemic.

AIMS

The primary aim of the study is:

To describe the incidence of HIV and other STIs during the study period.

The specific aims of the study are:

To provide harm reduction through clinical follow-up for informal PrEP users. To describe the conditions of informal use and acquisition of PrEP. To evaluate the effectiveness and safety of informal PrEP. To describe the demographic, clinical, risk factors for HIV and other STIs of informal PrEP users.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 yo at the time of the enrollment in the study.
* Accept voluntarily participation through signing informed consent, once explained its characteristics.
* Have obtained recently (less than 1 month) a negative result in the combined antigen/antibody rapid test / 4th generation ELISA or PCR HIV test.
* Active user or intending to use informal PrEP.

Exclusion Criteria:

* People with known HIV diagnosis.
* Absolute contraindication (eg known hypersensitivity to the active ingredients FTC or TDF) of the use of PrEP.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is addressed to men who have sex with men and transgender women
Study Population: Potential participants will be those who report using or intend to use PrEP, attending the community centers on a regular or spontaneous basis. Potential participants may be recruited for the study if they meet all inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of HIV and other STIs during the study period. | 36 months

SECONDARY OUTCOMES:
Number of people / visits = Number of visits / people who attend any visit | 36 months
  This indicator will be calculated for both the number of visits and the number of people.
  Disaggregation: based on sociodemographic characteristics and type of visit and PrEP guidelines
Retention percentage in the program | 36 months
  % retention in the program = (People who complete the study as per protocol) / (People enrolled) x100 Disaggregation: based on sociodemographic characteristics, presence of other STIs, use of drugs and number of sexual partners.
Number of medicines-related problems | 36 months
  Number of problems = Number of medicines-related problems Disaggregation:based on type of problem as per protocol, sociodemographic characteristics, use of drugs, medication, way of acquisition and other relevant factors
Number of negative results of the medication | 36 months
  Number of negative results of the medication = Number of negative results of the medication Disaggregation: based on type of negative result as per protocol, sociodemographic characteristics, drug use, medication, way of acquisition and other relevant factors

CONTACTS AND LOCATIONS:
Overall Officials: Pep Coll, MD, Principal Investigator — Fundación Lucha contra el Sida
Locations (1):
- BCN Checkpoint, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website of BCN Checkpoint — http://www.bcncheckpoint.com/
- See also: website of Fundación Lucha contra el Sida — https://www.flsida.org/es